CLINICAL TRIAL: NCT05805956
Title: An Open-label, Multicenter, First-in-human Dose-escalation and Cohort Expansion Phase I/II Clinical Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of IMM2902 in the Treatment of HER2-expressing Advanced Solid Tumors
Brief Title: IMM2902 in Patients With Advanced Solid Tumors Expressing HER2
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMM2902-001
Record Dates: First submitted 2023-03-23; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumor; Advanced Lung Cancer; Advanced Gastric Carcinoma; Advanced Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IMM2902 (Experimental): Phase 1 is the dose escalation part, patients with HER2 expressing solid tumors will be enrolled in groups of different dose levels, to explore MTD, RP2D, safety, and preliminary efficacy of IMM2902.
  Phase 2 is the cohort expansion part, patients with HER2 overexpressing advanced solid tumors will be enrolled in three cohorts, to explore the safety and efficacy of IMM2902.
  Interventions: Drug: IMM2902

INTERVENTIONS:
Drug: IMM2902 — a recombinant bispecific monoclonal antibody with high affinity to the dual targets, HER2 and CD47

SUMMARY:
This trial is an open-label, multicenter, first-in-human dose-escalation and cohort expansion Phase I/II clinical study to evaluate the safety, tolerability and preliminary efficacy of IMM2902 in the treatment of HER2-expressing advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the Informed Consent Form (ICF) and follow the protocol requirements;
2. Age ≥ 18 years old and ≤ 75 years old, regardless of gender;
3. Expected survival time ≥ 12 weeks;
4. HER2 expression:

   HER2 protein expression or HER2 gene amplification was found in primary or metastatic tumor tissue (IHC) or FISH.

   Phase I (dose escalation phase):

   HER2 expression is defined as IHC1+, IHC2+ or IHC3+, FISH testing is not required, and testing results from local qualified medical institutions are acceptable.

   Phase II (cohort expansion phase):

   HER2 overexpression is defined as IHC 3+ or IHC 2+, which can be tested by local qualified medical institutions.
5. Clinical diagnosis:

   Phase I (dose escalation phase):

   Patients with advanced solid tumors with HER2 expression (IHC1+, IHC2+ or IHC3+) confirmed by histology or cytology, who have previously received standard treatment progress, treatment ineffective or no standard treatment plan, including but not limited to breast cancer, gastric cancer (including gastroesophageal combination adenocarcinoma), urothelial carcinoma, biliary tract carcinoma, ovarian cancer, colon cancer and non-small cell lung cancer.

   Phase II (cohort expansion phase), including 3 cohorts:

   Cohort 1: Histologically or cytologically confirmed unresectable locally advanced or metastatic non-small cell lung cancer with HER2 overexpression (IHC3+ or IHC2+), who have previously failed systemic therapy; Cohort 2: Unresectable locally advanced or metastatic gastric cancer (including gastroesophageal junction adenocarcinoma) with histologically or cytologically confirmed HER2 overexpression (IHC3+ or IHC2+), who have previously received at least two systemic regimens.

   Cohort 3: Unresectable locally advanced or metastatic biliary tract cancer with histologically or cytologically confirmed HER2 overexpression (IHC3+ or IHC2+), recurrence or disease progression after previous standard treatment.
6. Patients included in the Phase II study need to provide previous HER2 test results, or archive tumor tissue to detect HER2 expression status. If neither is available, the patient may undergo a new tumor biopsy.
7. According to the evaluation criteria for solid tumors (RECIST v1.1), measurable lesions (longest diameter of spiral CT scan ≥ 10 mm, if the lesion is a lymph node, the short axis ≥ 15 mm; and the lesion has not received radiotherapy, unless the lesion clear progress); Phase I (dose escalation phase): Evaluable lesions (target lesions or non-target lesions); Phase II (Cohort Expansion Phase): Measurable lesions (target lesions) according to RECIST v1.1 criteria.
8. Eastern Cooperative Oncology Group (ECOG) score 0 or 1;
9. Adequate organ and coagulation function
10. AE related to previous systemic chemotherapy, radical/extensive radiotherapy or other antineoplastic drug treatment recovered to (NCI CTCAE v5.0)≤ Grade 1 (except for non-clinically significant or asymptomatic laboratory abnormalities), Patients with controlled grade 2 hypothyroidism and hyperglycemia may be enrolled after consultation with the sponsor;
11. Cumulative dose of anthracycline doxorubicin ≤360mg/m2 or its equivalent dose, epirubicin ≤720mg/m2;

10. Patients of childbearing age must take effective contraceptive measures during the study to within 6 months after the last dose.

Exclusion Criteria:

1. Received the last systemic or local anti-tumor therapy within 4 weeks before the first administration, including chemotherapy, immunotherapy, biological agents, etc.; received hormone anti-tumor therapy, small molecule targeted therapy within 2 weeks before the first administration; Palliative local treatment for non-target lesions within 2 weeks before the first administration; received non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, tumor necrosis factor, etc., not including IL-11 for the treatment of thrombocytopenia); Chinese herbal medicine or Chinese patent medicine with anti-tumor indications within 1 week before the first administration.
2. Received therapeutic drugs targeting SIRPα/CD47 4 weeks before the first administration, such as CD47 antibody, SIRPα fusion protein, SIRPα antibody and SIRPγ fusion protein;
3. Patients with primary central nervous system (CNS) malignant tumors or active CNS metastases who have failed local treatment (radiotherapy or surgery), but the following patients are allowed to enroll: a. Asymptomatic brain metastases; b. Clinical symptoms are stable (that is, there is no imaging progress 4 weeks before the first administration, and any neurological symptoms have returned to the baseline level), and corticosteroids and other treatments for brain metastases are not required for ≥4 weeks;
4. Uncontrolled hypertension (systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg) or pulmonary hypertension or unstable angina pectoris; myocardial infarction or bypass or stent surgery within 6 months before administration; Chronic heart failure history of grade III-IV of NYHA criteria; clinically significant valvular disease; serious arrhythmia requiring treatment (except atrial fibrillation, paroxysmal supraventricular tachycardia), including male QTc ≥ 450ms, Female QTc≥470ms (calculated by Fridericia formula); cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 12 months before enrollment;
5. History of arterial thrombosis, deep vein thrombosis and pulmonary embolism within 3 months before the first administration;
6. Have a history of moderate or severe dyspnea at rest due to advanced malignant tumors or their complications or severe primary lung diseases, or currently require continuous oxygen therapy, or currently suffer from interstitial lung disease (ILD), severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc.;
7. Suffering from other malignant tumors within 5 years before the first administration. Except: a. Cervical carcinoma in situ or non-melanoma skin cancer that has been radically cured; b. Second primary cancer that has been radically cured and has no recurrence within five years; c. The investigators believe that both primary cancers can benefit from this study;
8. Diseases that may cause gastrointestinal bleeding or perforation (such as duodenal ulcer, intestinal obstruction, acute Crohn's disease, ulcerative colitis, large-scale gastric and small intestinal resection, etc.); patients with chronic Crohn's disease and patients with ulcerative colitis (except those with total colon and rectal resection), even in the inactive phase, should be excluded; those with hereditary nonpolyposis colorectal cancer or familial adenomatous polyposis syndrome; Perforation, intestinal fistula history, but not cured after surgical treatment; esophageal and gastric varices;
9. Need puncture and drainage to treat uncontrollable pleural, abdominal and pericardial effusions that require repeated drainage or have obvious symptoms;
10. Have active hepatitis B [hepatitis B virus surface antigen (HBsAg) positive and/or hepatitis B virus antibody (HBcAb) positive, and HBV DNA ≥ 2000 IU/ml, and hepatitis caused by drugs or other reasons is excluded], or active hepatitis C [anti-hepatitis C virus (HCV) antibody positive, and HCV RNA is higher than the lower limit of detection, and hepatitis caused by drugs or other causes is excluded];
11. Has a history of immunodeficiency, including human immunodeficiency virus (HIV) infection, or other immunodeficiency diseases, or has a history of organ transplantation;
12. Have a history of autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, autoimmune thyroid disease, multiple sclerosis, etc. patient. except:

    1. Hypothyroidism that can be controlled only by hormone replacement therapy;
    2. Skin diseases that do not require systemic treatment (such as vitiligo, and psoriasis);
    3. Controlled celiac disease. However, patients who are using immunosuppressants or systemic hormone therapy (prednisone or other equivalent hormones at a dose ≥ 10 mg/day) and continue to use them within 2 weeks before enrollment cannot be enrolled;
13. Evidence of uncontrollable severe active infection (such as sepsis, bacteremia, viremia, etc.);
14. Have a history of allergies of grade 3 or above to any component or excipient of the study drug; or have a history of allergic reactions of grade 3 or above to trastuzumab or other anti-HER2 targeted drugs (CTCAE v5.0 classification);
15. Received anti-tumor vaccine treatment 4 weeks before the first administration or plan to receive anti-tumor vaccine trial;
16. Have undergone major surgery within 4 weeks before the first administration and have not fully recovered, or plan to undergo major surgery in the first 12 weeks after receiving the study drug; have received minor surgery (including catheterization) 2 days before enrollment, except for central venous catheterization via peripheral venipuncture);
17. Those who have a clear history of neurological or mental disorders, such as epilepsy, dementia, and poor compliance;
18. Has a history of alcoholism or drug abuse in the past 1 year;
19. Serum pregnancy test positive or breastfeeding women; do not agree to take adequate contraceptive measures during the study period and within 6 months after receiving the test drug;
20. Patients who have participated in other clinical studies in the past shall be out of the group in accordance with original clinical studies and more than 4 weeks prior to the first administration of this study;
21. Other situations where investigators believe they are inappropriate for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) of IMM2902 | 48 weeks
  Observe the safety and tolerability of IMM2902 in patients with advanced solid tumors expressing human epidermal growth factor receptor 2 (HER2), so as to determine the MTD
recommended phase 2 dose (RP2D) of IMM2902 | 48 weeks
  Observe the safety and tolerability of IMM2902 in patients with advanced solid tumors expressing human epidermal growth factor receptor 2 (HER2), so as to determine the RP2D
Treatment-related adverse events as assessed by CTCAE v5.0 | 48 weeks
  To evaluate the safety of IMM2902
objective response rate | 48 weeks
  proportion of subjects whose tumors achieved CR and PR after treatment
disease control rate | 48 weeks
  the proportion of subjects whose tumors achieved CR, PR and SD after treatment
duration of response | 48 weeks
  the time from the beginning of recording an objective response to the first occurrence of tumor progression, or death from any cause
progression-free survival | 48 weeks
  the time from the start of treatment to tumor progression or death from any cause

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - 301 Hospital, Beijing
  - Fudan University Cancer Hospital, Shanghai